CLINICAL TRIAL: NCT06165354
Title: Evaluating the Effectiveness in Supportive Treatment of Vaginitis of Vaginal-spraying Bacillus Probiotic Spore Suspension (LiveSpo X-Secret)
Brief Title: Effects of LiveSpo X-SECRET in SupportiveTreatment of Vaginitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anabio R&D (Industry)
Collaborators: Hanoi Obstetrics and Gynecology Hospital (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TNLS.2023.X; CS/PSHN/DC/23/38 (Other: Hanoi Obstetrics and Gynecology Hospital)
Record Dates: First submitted 2023-11-22; First posted 2023-12-11 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Vaginitis
Keywords: Bacterial vaginosis (BV); Sexually Transmitted Diseases (STDs); Vaginal-spraying probiotics; Bacillus spores; Bacteria; Fungi; Virus; Vietnamese women
MeSH Terms: conditions — Vaginitis; Vaginosis, Bacterial; Sexually Transmitted Diseases; Virus Diseases

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Parallel Assignment Blind, randomized, and controlled clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: LiveSpo X-secret and placebo 0.9% NaCl physiological saline are indistinguishable regarding taste and smell. The color and turbidity of LiveSpo X-secret suspension is unrecognizable to investigators except the PI and analyzer due to opaque plastic container.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator): Control group receives the routine treatment and uses 0.9% NaCl physiological saline.
  The routine treatment regimen at Hanoi Obstetrics and Gynecology Hospital (Hanoi OGH) and Bac Ninh Center for Disease Control and Prevention (Bac Ninh CDC) depends on clinical symptoms, test results of bacterial staining and pathogen detected using multiplex real time PCR assay on day 0.
  Interventions: Drug: 0.9% NaCl physiological saline
- X-secret (Experimental): X-SECRET group receives the routine treatment and uses NaCl 0.9% plus B. subtilis, B. clausii, and B. coagulans at 5 billion CFU/5 mL (LiveSpo®️ X-SECRET).
  The routine treatment regimen at Hanoi OGH and Bac Ninh CDC depends on clinical symptoms, test results of bacterial staining and pathogen detected using multiplex real time PCR assay on day 0.
  Interventions: Combination Product: LiveSpo X-secret

INTERVENTIONS:
Drug: 0.9% NaCl physiological saline — Vaginal-spraying 0.9% NaCl physiological saline is prepared by extracting 10 mL from 0.9% NaCl intravenous infusion 500 mL PP bottle (B.Braun, Germany, product declaration No. VD-32732-19), and then pouring it into the same opaque metallic spraying 20 mL-bottle.
  Other Names: Registration number: VD-32723-19
  Arms: Control
Combination Product: LiveSpo X-secret — In Vietnam, LiveSpo X-SECRET is manufactured as two product lines: (1) Class-A medical device product (Product declaration No.220003286/PCBA-HN) under manufacturing standards approved by Hanoi Department of Health, Ministry of Health, Vietnam and ISO 13485:2016 (Certificate No YT117-19) and (2) comestic (Product declaration No.14981/22/CBMP-HA) under manufacturing standards approved by Hanoi Department of Health, Ministry of Health, Vietnam (Certificate No 118/CNĐĐKSXMP. Both product lines have the same probiotic composition.
  The cosmetic type was used for the clinical trial conducted at Hanoi OGH. The Class-A medical device type was used for the clinical trial conducted at Bac Ninh CDC.
  Other Names: Registration number: No.220003286/PCBA-HN; Registration number: 14981/22/CBMP-HA
  Arms: X-secret

SUMMARY:
Vaginitis is a common reproductive infection in women worldwide, particularly in tropical and underdeveloped countries. Traditional antibiotic treatments can disrupt the balance of beneficial bacteria, requiring repeated use, seriously affecting women's health. Therefore, probiotics are microorganisms that are beneficial to human health when consumed in sufficient amounts, playing an important role in maintaining the balance of the body's microflora, especially in the intestines and vagina. Many studies around the world have proven that probiotic strains belonging to the genera Lactobacillus, Bifidobacterium, Bacillus, and Saccharomyces can help reduce the incidence and severity of bacterial vaginal infections and yeast infections. However, the effectiveness of oral or tablet probiotics is limited due to a slow onset of action and sensitivity to acidic conditions and temperature. In this study, the investigators proposed that vaginal spray probiotics containing Bacillus strains combined with proven stability in both acidic and thermal environments, may be a safe and effective symptomatic treatment for vaginal infections due to pathogenic bacteria, viruses, fungi, and/or flagellates. This probiotic supportive therapy may offer a promising alternative to traditional antibiotic therapy by (i) inhibiting the growth of pathogenic microorganism; (ii) regulating pro-inflammatory cytokines; and (iii) improving vaginal microbiota.

The aim of the study is to evaluate the effectiveness of vaginal-spraying Bacillus probiotics in LiveSpo®️ X-SECRET (5 billion CFU/5 mL B. subtilis, B. clausii, and B. coagulans) in preventing and supporting the treatment of vaginal infections.

Study Population: The study is being carried out at Hanoi Obstetrics and Gynecology Hospital (Hanoi OGH) and Bac Ninh Center for Disease Control and Prevention (Bac Ninh CDC). The sample size is 120 per each location.

Description of Study Intervention: In each location, a total of 120 eligible patients are recruited and divided randomly into 2 groups (n = 60/group/location): Control and Experimental groups. Patients in the Control group received routine treatment and 2-3 times/day 0.9% NaCl physiological saline while patients in the experimental group were treated with LiveSpo X-SECRET 2-3 times/day in addition to the same standard of care treatment. While the standard treatment regimen lasts for 7 days, the probiotic treatment is continually maintained for 28 days.

Study duration: 8 months.

DETAILED DESCRIPTION:
Vaginitis is a disease related to women's reproductive tract including bacterial vaginosis (Bacterial vaginosis - BV), sexually transmitted diseases (Sexually Transmitted Diseases - STDs)... This is considered is a common infection in the world, especially in developing and underdeveloped tropical countries, with up to 3/4 of the population suffering from STDs, mainly in the reproductive age group of 15-24. There are many microbial agents that cause gynecological diseases, including bacteria, viruses, fungi, flagellates... Bacterial vaginosis is an endogenous vaginal infection caused by more than 30 different species of bacteria, mainly mainly anaerobic bacteria such as Gardnerella vaginalis, Mycoplasma hominis, M. genitalium... Vaginitis is quite common in Vietnamese women. This is an issue of great concern in public health care because sexually transmitted diseases often have mild or no symptoms, so they are easy to ignore. Besides, the use of broad-spectrum antibiotics can lead to side effects such as loss of appetite, fatigue and sexual problems, while repeated treatments can lead to the appearance of antibiotic resistance, poses a significant challenge to the treatment of BV and STDs worldwide. The disease is normally caused by the replacement of Lactobacillus (a group of beneficial bacteria of the vagina) leading to an overgrowth of anaerobic bacteria. Probiotics are microorganisms that are beneficial to human health when consumed in sufficient amounts, playing an important role in maintaining the balance of the body's microflora, especially in the intestines and vagina. Studies have found that probiotics may help reduce the incidence and severity of vaginal infections, including bacterial vaginosis and yeast infections. Currently, probiotics formulated as oral capsules or gynecological suppositories containing Bifidobacterium or Lactobacillus strains are being studied as a potential adjunctive therapy for the treatment of vaginal infections. However, these strains have low viability and are sensitive to temperature, humidity and pH, making preservation difficult. Their effectiveness therefore depends on the specific strains used and the dosage required to achieve high concentrations in the vaginal tract. Beneficial bacteria of the Bacillus genus have been studied for a long time for their safety. For example, Bacillus subtilis, B. clausii and B. coagulans are often aerobic or facultative anaerobic bacteria, capable of growing rapidly and forming spores that are resistant to harsh conditions such as lack of nutrition, lack of oxygen, high temperatures and even antibiotics. In addition, these bacteria are particularly well-suited for usage as direct and in-situ probiotic vaginal sprays since they can also secrete antibacterial compounds, lactic acid, H2O2, and activate the mucosal layer of intestinal immune system. The vaginal-spraying probiotic therapy helps support the treatment and prevention of sexually transmitted pathogens, providing a promising support/alternative solution to traditional antibiotic therapy.

The aim of this study is to assess if vaginal-spraying Bacillus probiotic spores can can reduce clinical symptoms and improve various sub-clinical markers of vaginitis patients.

Methods: Prospective design of randomized, double-blind, and controlled clinical trial. The experiment was conducted on women with vaginitis and the obtained data was compared either between 2 groups or among two-to-four time points of treatment period of the same group. The control group was applied the routine treatment at the hospital combined with spraying 0.9% NaCl physiological saline into the vagina 3 times/time x 2 times/day continuously for 28 days. The test group was applied routine treatment at the hospital combined with spraying LiveSpo X-SECRET into the vagina 3 times/time x 2 times/day continuously for 28 days.

Samples are taken at day 0 and one or more of the following time points: day 3, 7, 14, and/or 28, depending on each research unit's ability to control sampling at certain intervals during the treatment procedure. In details, samples were taken at day 0, 7, and 28 at Hanoi OGH; and at day 0, 3, 7, 14, 28 at Bac Ninh CDC. Sub-clinical indicators related to vaginitis was monitored at different time points, including:

* Bacterial staining tests: These tests were conducted routinely at the Departments of Microbiology, both at Hanoi OGH and Bac Ninh CDC, at day 0 and day 28.
* Real time PCR assay to detect 9 main microorganisms that cause inflammation in vaginal swab samples: Gardnerella vaginalis (GV); Neisseria gonorrhoeae (NG); Chlamydia trachomatis (CT); Candida albicans (CA); Trichomonas vaginalis (TV); Mycoplasma hominis (MH); Mycoplasma genitalium (MG); Human alphaherpesvirus type 1 (HSV-1); Human alphaherpesvirus type 2 (HSV-2). This assay was performed at the Department of Microbiology, Fungi, and Parasitology Testing, Central Dermatology Hospital, using commercial kits or an "in-house" kit that was recently developed and published internationally by the research team (Bui et al. ., 2023). The assay was carried out at day 0, 7, and 28 for samples collected at Hanoi OGH; and at day 0, 3, 7, 14, 28 for samples collected at Bac Ninh CDC.
* Real time PCR assay to detect Bacillus sp. including B. subtilis, B. clausii and B. coagulans in vaginal swab samples. This experiment was performed at the Spobio Research Center, Anabio R&D. The assay was carried out at day 0, 7, and 28 for samples collected at Hanoi OGH; and at day 0, 3, 7, 14, 28 for samples collected at Bac Ninh CDC.
* Analysis of immune index including 5 types of cytokines IL-1β, IL-6, IL-8, IL-10, TNF-α and IgA was performed using ELISA technique from vaginal swab samples collected at days 0, 7, and 28 at Hanoi OGH only. The tests are conducted at the Department of Microbiology, Fungi, and Parasitology Testing, Central Dermatology Hospital or Spobio Research Center, Anabio R&D.
* Changes in microbiome using 16S rRNA metagenome analysis: This microbiome analysis was conducted for representative vaginal swab samples from patients of each research group (expected 10-15 patients/group) using new generation sequencing (NGS) on an Illumina MiSeq system (Illumina, San Diego, CA, USA) with a 2 × 250 bp run configuration. The assay was carried out at day 0 and one or more of the following time points day 7 and 28 for samples collected at both Hanoi OGH and Bac Ninh CDC.

ELIGIBILITY:
Inclusion Criteria:

* Women from 18 to 60 years old
* Diagnosed with vaginitis with obvious symptoms and manifestations such as: vulvar/vaginal ulcers, inflammation, vaginal odor, vaginal itching, vaginal cololr, painful/ painful urination, lower abdominal pain; pain during sex; abnormal vaginal bleeding…
* Positive for one of the following pathogents that cause vaginitis, such as Gardnerella vaginalis, Mycoplasma hominis, Candida albicans, Chlamydia trachomatis, Neisseria gonorrhoeae, Mycoplasma genitalium, HSV-1, HSV-2, Trichomonas vaginalis, detected by real-time PCR assay.
* The patient agrees to participate in the study, explains and signs the consent form to participate in the study.

Exclusion Criteria:

* Women who are pregnant or breast-feeding, have diabetes, are using antibiotics/anti-inflammatory drugs in the vaginal area within the previous 14 days
* Vaginal bleeding of unknown cause or cancer
* Have a history of drug allergy and hypersensitivity to any ingredient in probiotics or placebo
* Leave the study before day 7
* Simultaneous participation in another clinical trial or use of probiotics for the gynecological tract within the past 14 days
* Meets criteria for mental, cognitive, depressive or anxiety disorders
* Do not agree to participate in the study

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Vagninitis infection in women.
Enrollment: 120 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with free and/or reduced gynecological infection symptoms | Day 0, 3, 7, 14, and 28
  Vulvar and vaginal ulcers (rating from 0 to 3 on a scale of: no ulcers - 0, labia minora ulcers, small, no pain-1, larger or painful ulcer - 2, very large, painful and rapidly spreading ulcer - 3) Inflammation (rating from 0 to 3 on a scale of: none - 0, mild redness or inflammation - 1, swelling or pain in vulva, vagina, or groin - 2, swollen lymph nodes and groin pain - 3) Itching (rating from 0 to 3 on a scale of: none - 0, mild itching or irritation - 1, itching, burning - 2, severe and persistent itching, burning - 3) Vaginal fluid color (uniform-clear white - 0, opalescent white - 1A, yellow/green - 1B; grey white - 1C) Vaginal odor (No/Yes) Painful/ painful urination (No/Yes) Lower abdominal pain (No/Yes) Abnormal vaginal bleeding (No/Yes)

SECONDARY OUTCOMES:
Changes in the vaginal pathogens load | Day 0, 3, 7, 14, and 28
  Changes in the load or concentration of pathogens in vaginal samples, as indicated by real-time PCR threshold cycle (Ct) value at one or more of the following time points: day 3, 7, 14 and/or day 28 (after treatment) compared to day 0 (before treatment).
Changes in immune indices in vaginal samples before and after treatment | Day 0, 3, 7, 14, and 28
  Vaginal mucosal cytokines (pg/mL) including: interleukin-1β (IL-1β), interleukin-6 (IL-6), interleukin-8 (IL-8), interleukin-10 (IL-10), tumor necrosis factor-α TNF-α
  Vaginal mucosal (µg/mL) pro-inflammatory IgA.
Changes in other patient's sub-clinical indicators in vaginal samples before and after treatment | Day 0, 3, 7, 14, and 28
  * Clue cells (Negative/Positive)
  * Neisseria gonorrhoeae (Negative/Positive)
  * Fungi (Negative/Positive)
  * Trichomonas (Negative/Positive)
  * Vaginal epithelial cells (Negative/Positive)
Changes in vaginal microbiota vaginal samples before and after treatment | Day 0,7, and 28
  Composition (diversity and abundance) of phylum, family, genus, and species of vaginal samples was analysed based on the data of 16S rRNA metagenome using next-generation sequencing (NGS). The analysis was carried out at day 7 or/ and day 28 (after treatment) compared with day 0 (before treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Chuong C Nguyen, MSc. MD, Principal Investigator — Hanoi Obstetrics and Gynecology Hospital; Anh TV Nguyen, Assoc. Prof., Principal Investigator — Spobio Research Center, Anabio R&D; Thuy TB Nguyen, MSc. MD, Principal Investigator — Hanoi Obstetrics and Gynecology Hospital; Ngoc TB Nguyen, MD, Principal Investigator — Hanoi Obstetrics and Gynecology Hospital; Hong T Ngo, MSc, Principal Investigator — Bac Ninh Center for Disease Control and Prevention; Huyen T Bui, Principal Investigator — Spobio Research Center, Anabio R&D; Hao TN Vo, Principal Investigator — Spobio Research Center, Anabio R&D
Locations (2):
- Vietnam (2):
  - Centers for Disease Control and Prevention, Bắc Ninh, Bac Ninh
  - Hanoi Obstetrics and Gynecology Hospital, Ba Dinh, Hanoi

IPD SHARING:
Plan to Share IPD: Yes
Data or samples share that will be coded, with no PHI include. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research and will be provided following review and approval of a study protocol, informed consent form (ICF), clinical study peport (CSR). For more information or to submit a request, please contact anabio.rd2021@gmail.com

REFERENCES:
- [Background] Izetbegovic S, Alajbegovic J, Mutevelic A, Pasagic A, Masic I. Prevention of diseases in gynecology. Int J Prev Med. 2013 Dec;4(12):1347-58. PMID 24498489
- [Background] Morrill S, Gilbert NM, Lewis AL. Gardnerella vaginalis as a Cause of Bacterial Vaginosis: Appraisal of the Evidence From in vivo Models. Front Cell Infect Microbiol. 2020 Apr 24;10:168. doi: 10.3389/fcimb.2020.00168. eCollection 2020. PMID 32391287
- [Background] Peebles K, Velloza J, Balkus JE, McClelland RS, Barnabas RV. High Global Burden and Costs of Bacterial Vaginosis: A Systematic Review and Meta-Analysis. Sex Transm Dis. 2019 May;46(5):304-311. doi: 10.1097/OLQ.0000000000000972. PMID 30624309
- [Background] Le T, Kinh NV, Cuc NTK, Tung NLN, Lam NT, Thuy PTT, Cuong DD, Phuc PTH, Vinh VH, Hanh DTH, Tam VV, Thanh NT, Thuy TP, Hang NT, Long HB, Nhan HT, Wertheim HFL, Merson L, Shikuma C, Day JN, Chau NVV, Farrar J, Thwaites G, Wolbers M; IVAP Investigators. A Trial of Itraconazole or Amphotericin B for HIV-Associated Talaromycosis. N Engl J Med. 2017 Jun 15;376(24):2329-2340. doi: 10.1056/NEJMoa1613306. PMID 28614691
- [Background] Tuddenham S, Hamill MM, Ghanem KG. Diagnosis and Treatment of Sexually Transmitted Infections: A Review. JAMA. 2022 Jan 11;327(2):161-172. doi: 10.1001/jama.2021.23487. PMID 35015033
- [Background] Ton Nu PA, Nguyen VQ, Cao NT, Dessi D, Rappelli P, Fiori PL. Prevalence of Trichomonas vaginalis infection in symptomatic and asymptomatic women in Central Vietnam. J Infect Dev Ctries. 2015 Jul 4;9(6):655-60. doi: 10.3855/jidc.7190. PMID 26142677
- [Background] Mastromarino P, Macchia S, Meggiorini L, Trinchieri V, Mosca L, Perluigi M, Midulla C. Effectiveness of Lactobacillus-containing vaginal tablets in the treatment of symptomatic bacterial vaginosis. Clin Microbiol Infect. 2009 Jan;15(1):67-74. doi: 10.1111/j.1469-0691.2008.02112.x. Epub 2008 Nov 22. PMID 19046169
- [Background] de Boer AS, Diderichsen B. On the safety of Bacillus subtilis and B. amyloliquefaciens: a review. Appl Microbiol Biotechnol. 1991 Oct;36(1):1-4. doi: 10.1007/BF00164689. No abstract available. PMID 1367772
- [Background] Ratna Sudha M, Yelikar KA, Deshpande S. Clinical Study of Bacillus coagulans Unique IS-2 (ATCC PTA-11748) in the Treatment of Patients with Bacterial Vaginosis. Indian J Microbiol. 2012 Sep;52(3):396-9. doi: 10.1007/s12088-011-0233-z. Epub 2011 Sep 23. PMID 23997330
- [Background] Tsimaris P, Giannouli A, Tzouma C, Athanasopoulos N, Creatsas G, Deligeoroglou E. Alleviation of vulvovaginitis symptoms: can probiotics lead the treatment plan? Benef Microbes. 2019 Dec 9;10(8):867-872. doi: 10.3920/BM2019.0048. PMID 31965832
- [Background] Lee NK, Kim WS, Paik HD. Bacillus strains as human probiotics: characterization, safety, microbiome, and probiotic carrier. Food Sci Biotechnol. 2019 Oct 8;28(5):1297-1305. doi: 10.1007/s10068-019-00691-9. eCollection 2019 Oct. PMID 31695928
- [Background] Li C, Wang T, Li Y, Zhang T, Wang Q, He J, Wang L, Li L, Yang N, Fang Y. Probiotics for the treatment of women with bacterial vaginosis: A systematic review and meta-analysis of randomized clinical trials. Eur J Pharmacol. 2019 Dec 1;864:172660. doi: 10.1016/j.ejphar.2019.172660. Epub 2019 Sep 25. PMID 31562865
- [Background] Bui HTV, Bui HT, Chu SV, Nguyen HT, Nguyen ATV, Truong PT, Dang TTH, Nguyen ATV. Simultaneous real-time PCR detection of nine prevalent sexually transmitted infections using a predesigned double-quenched TaqMan probe panel. PLoS One. 2023 Mar 6;18(3):e0282439. doi: 10.1371/journal.pone.0282439. eCollection 2023. PMID 36877694
- [Derived] Bui HT, Bui ATP, Ngo HT, Ngo XT, Nguyen HT, Nguyen AH, Tran VC, Pham TD, Nguyen ATV. Vaginal-spray Bacillus spore probiotics as a potential treatment and reducing recurrence of bacterial vaginosis: randomized, double-blind, and controlled pilot study. Commun Med (Lond). 2025 Nov 18;5(1):527. doi: 10.1038/s43856-025-01236-4. PMID 41258468